CLINICAL TRIAL: NCT05624255
Title: Correlating the Measure of Retinal Vascular Density Through Angio-OCT with Calcium Score
Acronym: ANOSCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022/701
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Cardiovascular Abnormalities; Vascular Diseases; Retinal Vascular
MeSH Terms: conditions — Cardiovascular Abnormalities; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ophthalmology consultation (Experimental): Patients eligible to calcium score will be offered an ophthalmologic consultation including Angio-Optical Coherence Tomography [OCT]
  Interventions: Other: Ophthalmologic consultation

INTERVENTIONS:
Other: Ophthalmologic consultation — Complete ophthalmologic examination including angio-OCT

SUMMARY:
Recent case-control studies have proven that the retinal vascularization mirrors the cardiac vascularization: more the coronary network is altered, more the density of retinal vessels is reduced. No studies have yet been realised in primary prevention. This study aims to demonstrate a link between the density of the retinal vascularization and the calcium score, which is currently the gold standard for the classification of cardiovascular risk in primary prevention. Thus, a simple image of the retinal vascularization could predict the cardiovascular risk of a patient. OCT angiography would become a major aid in the classification of cardiovascular risk in asymptomatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for a calcium score as part of their standard treatment and volunteers for an ophthalmologic consultation

Exclusion Criteria:

* Pregnant women

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Correlation between retinal vascular density and calcium score | Day 1
  Comparison between values of calcium score and presence of vascular abnormalities in retina.
  Calcium is scored as follows:
  * Coronary Artery Calcium [CAC] = 0 : very low risk
  * CAC = [1-100[ : low risk
  * CAC = [100-400[ : moderate risque
  * CAC = [400-1000[ : high risk
  * CAC = > 1000 : very high risk

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No